CLINICAL TRIAL: NCT04687436
Title: Foley Catheter Versus Double-balloon Catheter for Cervical Ripening in Women With a High-risk Pregnancy
Brief Title: Foley Catheter Versus Double-balloon Catheter for Cervical Ripening
Status: Completed | Type: Observational
Sponsor: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Kemal Sarsmaz, Principal Investigator, Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Other Study IDs: mechanical cervical ripening
Record Dates: First submitted 2020-12-21; First posted 2020-12-29 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Cervical Ripening; Pregnancy, High-Risk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Foley catheter group: mechanical cervical ripening
  Interventions: Device: mechanical cervical ripening
- Double-balloon group: mechanical cervical ripening
  Interventions: Device: mechanical cervical ripening
- Cook cervical ripening balloon: mechanical cervical ripening
  Interventions: Device: mechanical cervical ripening

INTERVENTIONS:
Device: mechanical cervical ripening — mechanical cervical ripening with a foley catheter or double-balloon catheter or Cook cervical ripening balloon

SUMMARY:
The objective of this study is to compare pregnancy results which were used foley catheter or double-balloon catheter for cervical ripening among high-risk pregnant women.

DETAILED DESCRIPTION:
This is a prospective observational study. The planned sample size was calculated as 109 patients per group with 80% power and 0.05 alpha error.

The inclusion criteria are age between 18 and 40, singleton pregnancy, vertex presentation, bishop score <6, using a foley catheter or cook balloon for cervical ripening and high-risk pregnancy (Oligohydramnios, polyhydramnios, intrauterine growth retardation, pregestational or gestational diabetes, hypertensive disorders).

The exclusion criteria are being younger than 18 or over 40, communication problems, bishop score >6, being at active labor, multifetal pregnancy, non-vertex presentation, scarred uterus (cesarean or myomectomy), fetal structural or chromosomal anomaly, non-reassuring fetal cardiotocography before cervical ripening, regional anesthesia during the first stage.

The primary outcomes are the rate of bishop score >6 after ripening, vaginal delivery rate and vaginal delivery within 24 hours of the initiation of ripening.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40
* Singleton pregnancy
* Vertex presentation
* Bishop score <6
* Using a Foley catheter or cook balloon for cervical ripening
* High-risk pregnancy (Oligohydramnios, polyhydramnios, intrauterine growth retardation, pregestational or gestational diabetes, hypertensive disorders)

Exclusion Criteria:

* Being younger than 18 or over 40
* Communication problems (foreign national)
* Bishop score >6
* Being at active labor
* Multifetal pregnancy
* Non-vertex presentation
* Scarred uterus (cesarean or myomectomy)
* Fetal structural or chromosomal anomaly
* Non-reassuring fetal cardiotocography before cervical ripening
* Regional anesthesia during the first stage

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women with unfavorable cervices and need to deliver for maternal or fetal health condition.
Sampling Method: Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
bishop score | at the time of removing the cervical ripening catheter or when the balloon was expelled spontaneously
  bishop score >6 is accepted as successful ripening. (max. 10, and the higher bishop score means better ripening has been occurred.)
vaginal delivery rate | until the patient gives birth
  the difference in vaginal birth rate between groups
vaginal delivery within 24 hours | from the time of cervical ripening catheter insertion to the 24 hours
  the difference in vaginal delivery within 24 hours rate between groups

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Etlik Zubeyde Hanim Women's Health Care, Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Pennell CE, Henderson JJ, O'Neill MJ, McChlery S, Doherty DA, Dickinson JE. Induction of labour in nulliparous women with an unfavourable cervix: a randomised controlled trial comparing double and single balloon catheters and PGE2 gel. BJOG. 2009 Oct;116(11):1443-52. doi: 10.1111/j.1471-0528.2009.02279.x. Epub 2009 Jul 28. PMID 19656148
- [Background] Sayed Ahmed WA, Ibrahim ZM, Ashor OE, Mohamed ML, Ahmed MR, Elshahat AM. Use of the Foley catheter versus a double balloon cervical ripening catheter in pre-induction cervical ripening in postdate primigravidae. J Obstet Gynaecol Res. 2016 Nov;42(11):1489-1494. doi: 10.1111/jog.13086. Epub 2016 Jul 19. PMID 27436681